CLINICAL TRIAL: NCT06403319
Title: Otitis Media With Effusion Among Patients With Type 2 Inflammation Diseases
Brief Title: Otitis Media With Effusion and Type 2 Inflammation Diseases
Status: Completed | Type: Observational
Sponsor: Hearing and Language Healthcare Center, China Medical University Hsinchu Hospital, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: OME-S-24-00723
Record Dates: First submitted 2024-05-01; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Otitis media with effusion (OME) is thought to be associated with comorbidities such as allergic rhinitis, gastroesophageal reflux disease, asthma, and more. Many of these comorbidities can be caused by type 2 inflammation (T2I). This study aims to characterize the risk of undergoing OME surgery. This retrospective, matched-cohort study involved the retrospective recruitment of patients from 2009 to 2020, using the Taiwan National Health Insurance Research Database (NHIRD)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OME
* At least two outpatient visits or one hospitalization record
* Medical records within the database

Exclusion Criteria:

* Participants younger than 4 years old
* Participants with unclear demographic information
* Participants with a history of ear surgery or congenital ear anomalies
* Participants who had undergone OME surgery before the index date

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All study subjects with OME-confirmed by at least two outpatient visits or one hospitalization record within NHIRD database. We excluded cases that did not meet the following criteria: patients who had undergone OME surgery before the index date, individuals younger than 4 years old, patients with unknown demographic information, individuals in the comparison cohort with a history of T2I diseases, and patients with a history of ear surgery or congenital ear anomalies.
Sampling Method: Non-Probability Sample
Enrollment: 100622 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The number of participants with OME who requiring surgical intervention | 10 years
  surgical intervention including procedures such as myringotomy and adenoidectomy